CLINICAL TRIAL: NCT06267625
Title: Investigation of Dyspnea, Posture, Strength, Physical Activity, Functional Mobility and Balance in Elderly Individuals
Brief Title: Physical Impairments in Elderly Individuals
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Elderly Individuals
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Aging Disorder
Keywords: elderly individuals; older adults; dyspnea; posture; functional mobility; balance; muscle strength
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Individuals: This group will consist of individuals aged 65 and over
  Interventions: Other: Physical Evaluations of individuals

INTERVENTIONS:
Other: Physical Evaluations of individuals — Participants will be evaluated on posture, cough strength, functional mobility and hand grip strength.They will be asked to answer the Standardized Mini Mental Test, Modified Medical Research Council Scale, Physical Activity Scale for the Elderly, Berg Balance Scale. The data to be obtained from all these evaluations are planned to be collected face to face from the participants at once and within a maximum of 1 hour.

SUMMARY:
There are no studies in the literature reporting the dyspnea, posture, strength, physical activity, functional mobility and balance in elderly individuals. The aims of this observational study are; 1) to evaluate dyspnea, posture, strength, physical activity, functional mobility and balance in elderly individuals, 2) to reveal the relationships between these parameters of research group.

DETAILED DESCRIPTION:
The increase in the elderly population brings with it many health problems, especially in older ages. Rates of limitation and disability are increasing in elderly individuals due to chronic diseases. Many of these changes negatively affect their daily living activities. With aging, respiratory muscle strength and respiratory surface area decrease in the cardiopulmonary system. Respiration is negatively affected by the decrease in muscle strength. Postural correctness cannot be easily achieved in elderly individuals due to deterioration in bone, muscle and joint structures. Functional mobility and balance problems are observed with changes in postural control that occur with aging. There are not enough studies in the literature to clarify this issue that evalatues dyspnea, posture, strength, physical activity, functional mobility and balance in elderly individuals. Therefore, the aim of our study is to evaluate dyspnea, posture, strength, physical activity, functional mobility and balance in elderly individuals. Therefore, we aimed to clarify this gap.

ELIGIBILITY:
Inclusion Criteria for Elderly Individuals

* Being 65 years or older
* Volunteering to participate in the study
* Getting a score of 23 or higher on the Standardized Mini Mental State Test

Exclusion Criteria for Elderly Individuals

- The participant has a cognitive, neurological or orthopedic disease that would affect the participant's ability to move independently and understand the questions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: At least 50 individuals aged 65 and over will be included
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Dyspnea score | through study completion, an average of 1 year
  Dyspnea score will be obtained from the Modified Medical Research Council (MMRC) Scale. This scale is a five-item scale based on various physical activities that cause a feeling of shortness of breath (dyspnea). As the score an individual gets from the scale increases, the perception of shortness of breath also increases.

SECONDARY OUTCOMES:
Posture score | through study completion, an average of 1 year
  Posture deviation will be determined according to the deviation score in the joint centers obtained by photographing the posture of the individuals and uploading them to the system. Posture assessment will be made with a mobile application based on the concept of postural analysis with artificial intelligence.
Cough strength | through study completion, an average of 1 year
  Cough strength will be evaluated using a PEFmeter.
Handgrip strength | through study completion, an average of 1 year
  Hand grip strength will be measured using the Jamar hand dynamometer.
Functional mobility score | through study completion, an average of 1 year
  Functional mobility will be evaluated with Chair Stand Test. Higher repetition numbers indicate better physical performance.
Physical activity score | through study completion, an average of 1 year
  Physical activity will be assessed using the Physical Activity Scale for the Elderly. Participation in leisure activities, housework activities, and work-related activities are recorded. Higher score indicates better physical activity levels.
Functional Mobility score | through study completion, an average of 1 year
  Functional mobility and balance will be evaluated with Time Up and Go test. The test measures speed during many functional maneuvers such as standing, walking, turning and sitting.
Balance score | through study completion, an average of 1 year
  Balance will be assessed using Berg Balance Scale. The scale consists of 14 items. These items examine activities in which the support area gradually decreases and it becomes difficult to maintain the position.
Cognitive function score | through study completion, an average of 1 year
  Cognitive function will be assessed using the Standardized Mini Mental State Test. The maximum score is 30 points. Scores of 23 and lower indicate cognitive dysfunction, scores of 24 and above indicate normal cognitive level.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc.Dr, Study Director — Izmir Democracy University; ESRA SUDE AKIN, BSc, Principal Investigator — Izmir Democracy University; ÖZLEM ÇİNAR ÖZDEMİR, Assoc.Dr, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva CFR, Pegorari MS, Matos AP, Ohara DG. Dyspnea is associated with poor physical performance among community-dwelling older adults: a population-based cross-sectional study. Sao Paulo Med J. 2020 Mar;138(2):112-117. doi: 10.1590/1516-3180.2019.0428.R1.09122019. Epub 2020 Apr 9. PMID 32294715
- [Background] Dindorf C, Konradi J, Wolf C, Taetz B, Bleser G, Huthwelker J, Werthmann F, Bartaguiz E, Kniepert J, Drees P, Betz U, Frohlich M. Classification and Automated Interpretation of Spinal Posture Data Using a Pathology-Independent Classifier and Explainable Artificial Intelligence (XAI). Sensors (Basel). 2021 Sep 21;21(18):6323. doi: 10.3390/s21186323. PMID 34577530
- [Background] Kaulamo JT, Latti AM, Koskela HO. Recurrent Cough in the Elderly: A Forgotten Entity. Lung. 2023 Dec;201(6):545-553. doi: 10.1007/s00408-023-00654-2. Epub 2023 Nov 14. PMID 37964136